CLINICAL TRIAL: NCT00957229
Title: A Randomized, Phase II Multicenter Trial Evaluating the Efficacy and Safety of a Systemic Hedgehog Pathway Antagonist (GDC-0449) in Patients With Basal Cell Nevus Syndrome (BCNS)
Brief Title: To Determine The Efficacy and Safety of GDC-0449 in Patients With Basal Cell Nevus Syndrome (BCNS)
Acronym: GDC-0449
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-026; SHH-4685s (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2009-08-05; First posted 2009-08-12 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Basal Cell Nevus Syndrome; Gorlin Syndrome
MeSH Terms: conditions — Basal Cell Nevus Syndrome | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): placebo pill by mouth once daily
  Interventions: Drug: GDC-0449
- GDC-0449 (Experimental): vismodegib 150MG by mouth once daily
  Interventions: Drug: GDC-0449

INTERVENTIONS:
Drug: GDC-0449 — capsule, 150 mg, one pill daily, 18 months
  Other Names: Hedgehog Inhibitor; Hedgehog Antagonist

SUMMARY:
The purpose of this study is to reduce the number of new surgically eligible BCCs by 50% appearing during month 3-18 of medication ingestion.

DETAILED DESCRIPTION:
This is a Phase II, 18 month, double blind, randomized placebo-controlled, two arm multicenter clinical study design. During the 18-month treatment period, the safety and chemopreventive efficacy of 150 mg/day GDC-0449 versus placebo will be assessed, and include evaluations of the skin at monthly intervals for the first three months and then every 3 months for the next 15 months. Removal of new surgically eligible BCCs (SEBs) will be done by primary skin care physicians (PSCPs) or at Study Centers. A Data Safety Monitoring Board (DSMB) will review unblinded results for an interim analysis when 20 subjects have completed 12 months of drug. This review will focus on adverse events and efficacy results. Subjects will be monitored for the development of new SEBs after they discontinue study treatment. At the end of the 18 months, given that the observed adverse events are minimal, patients on placebo will be offered the opportunity to take GDC-0449 for 18 months in an open label continuation, followed by six months observation, and patients on GDC449 will be monitored for the next 24 months for assessment of the duration of benefit after stopping the drug.

ELIGIBILITY:
Inclusion Criteria:

The subject:

* has had diagnosed at least 10 SEB (of diameter 3 mm diameter or greater on the nose or periorbital skin, 5 mm or greater elsewhere on the face, or 9 mm or greater on non-facial areas excluding the skin below the knees) during the two years before study entry, as documented histologically in physicians' records and/or diagnosed clinically by a Study Investigator at baseline.
* meet diagnostic criteria for basal cell nevus syndrome
* is willing to abstain from application of non-study topical medications to the skin for the duration of the study, including prescription and over the counter preparations. Subjects will be encouraged to use sunscreen (SPF 15) at least once daily on all exposed skin sites.
* is willing to forego treatment of BCCs unless the BCCs are documented by Study Investigators, preferably on two separate visits, except when the PSCP believes that delay in treatment potentially might compromise the health of the subject.
* has normal laboratory tests as defined by the following: Normal hematopoietic capacity, Normal hepatic function: AST and ALT greater than or equal to 2x the upper limit of normal (ULN) Total bilirubin within normal range 0.20 mg/dl to 1.50 mg/dl or within 3x ULN for patients with Gilbert's disease Normal renal function: normal serum creatinine or measured creatinine clearance less than 50 mL/minute. Fasting cholesterol greater than or equal to 220 untreated
* be willing to not donate blood or semen for three months following discontinuation of Study medications.
* is willing to avoid pregnancy in his partner as defined by the following: Male subject is willing to use a latex condom during the study and for 3 months after the last dose during sexual contact with a female of childbearing potential, even if he has had a successful vasectomy. His partner must also use a form of birth control

Exclusion Criteria:

The subject:

* has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study. Specifically these include the use of: (i) glucocorticoids to more than 5% of the skin (ii) retinoids systemically or topically to more than 5% of the skin during the six months prior to study entry; (iii) alpha-hydroxy acids to more than 5% of the skin during the six months prior to study entry (iv) 5-fluorouracil or imiquimod systemically or topically to the skin above the knees during the six months prior to study entry. (v) treatment with systemic chemotherapy within one year prior to starting study medication.
* has a history of hypersensitivity to any of the ingredients in the study medication formulations.
* is unable to return for follow-up visits and tests.
* has uncontrolled systemic disease, including known HIV positive patients.
* has history of congestive heart failure.
* has uncontrolled hypocalcemia, hypomagnesemia, or hypokalemia
* has clinically important history of liver disease, including viral or hepatitis, current alcohol abuse, or cirrhosis.
* has any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study.
* has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or CLL Stage 0.
* has current, recent (within 4 weeks of Day 1), or planned participation in an experimental drug study while enrolled in this study.
* is a female who is pregnant, plans to ever to become pregnant, capable of becoming pregnant or is breast feeding.
* is a male who is unwilling or unable to comply with pregnancy prevention measures.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (2):
- United States (2):
  - Children's Hospital Oakland Research Institiute, Oakland, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang JY, Mackay-Wiggan JM, Aszterbaum M, Yauch RL, Lindgren J, Chang K, Coppola C, Chanana AM, Marji J, Bickers DR, Epstein EH Jr. Inhibiting the hedgehog pathway in patients with the basal-cell nevus syndrome. N Engl J Med. 2012 Jun 7;366(23):2180-8. doi: 10.1056/NEJMoa1113538. PMID 22670904
- [Result] Ally MS, Tang JY, Joseph T, Thompson B, Lindgren J, Raphael MA, Ulerio G, Chanana AM, Mackay-Wiggan JM, Bickers DR, Epstein EH Jr. The use of vismodegib to shrink keratocystic odontogenic tumors in patients with basal cell nevus syndrome. JAMA Dermatol. 2014 May;150(5):542-5. doi: 10.1001/jamadermatol.2013.7444. PMID 24623282
- [Result] Tang JY, Ally MS, Chanana AM, Mackay-Wiggan JM, Aszterbaum M, Lindgren JA, Ulerio G, Rezaee MR, Gildengorin G, Marji J, Clark C, Bickers DR, Epstein EH Jr. Inhibition of the hedgehog pathway in patients with basal-cell nevus syndrome: final results from the multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2016 Dec;17(12):1720-1731. doi: 10.1016/S1470-2045(16)30566-6. Epub 2016 Nov 10. PMID 27838224

RESULTS

PARTICIPANT FLOW:
Period: Study Start
Arm/Group | Sugar Pill | GDC-0449
Started | 15 | 26
Completed | 14 | 23
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Disease Progression | 1 | 0
Period: Reallocated to or Continued Vismodegib
Arm/Group | Sugar Pill | GDC-0449
Started | 14 | 23
Completed | 11 | 21
Not Completed | 3 | 2
Not completed — Death | 1 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | GDC-0449 | Total
Number analyzed (Participants) | 15 | 26 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (8) | 54 (8) | 54 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 18 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 26 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of New Surgically Eligible Basal-cell Carcinomas
Description: Number of new surgically eligible basal-cell carcinomas per patient per year
Time Frame: 3 months of receiving study drug
Measure: Mean (Standard Deviation); unit: events per patient year
Arm/Group | Sugar Pill | GDC-0449
Number analyzed (Participants) | 15 | 26
events per patient year | 34 (1.32) | 2 (0.12)

2. Secondary Outcome: Change in Size of the Existing Carcinomas, Expressed as the Sum of Cumulative Diameters in Millimeters Over an 18 Month Period
Time Frame: Baseline and 18 months
Measure: Number (95% Confidence Interval); unit: Millimeters
Arm/Group | Sugar Pill | GDC-0449
Number analyzed (Participants) | 15 | 26
Millimeters | 55 [NA to NA] — The PI has left the institution and the only access to the data is from the publication. The records no longer exist. All efforts have been made to obtain the data. | -60 [NA to NA] — The PI has left the institution and the only access to the data is from the publication. The records no longer exist. All efforts have been made to obtain the data.

3. Secondary Outcome: Number of New Surgically Eligible Basal-cell Carcinomas After Stopping Vismodegib Treatment
Description: The number of new surgically eligible basal-cell carcinomas per patient per month is reported.
Time Frame: These five patients were given placebo for a mean of 7.4 months (SD 2.3). After receiving vismodegib for a mean of 13.8 months (SD 6.8) and then discontinuing vismodegib for a mean of 11.8 months (SD 7.9) the new basal-cell carcinoma rate is reported.
Population: The incidence of new surgically eligible basal-cell carcinomas after stopping vismodegib was analysed in an exploratory analysis of the patients who crossed over to vismodegib and were followed up for at least 6 months after stopping vismodegib (n=5).
Measure: Mean (Standard Deviation); unit: carcinomas per patient per month
Arm/Group | Sugar Pill | GDC-0449
Number analyzed (Participants) | 5 | 5
carcinomas per patient per month | 1.7 (1.5) | 0.06 (0.12)

ADVERSE EVENTS:
Description: Grade 1 and 2 events are listed if considered related to vismodegib treatment. All other graded events are listed.
  The PI has left the institution and the only access to the data is from the publication, in which the data are reported as presented here. The records no longer exist. All efforts have been made to obtain the data.
Arm/Group | Sugar Pill | GDC-0449
All-Cause Mortality (participants affected / at risk) | 0/15 | 2/40
Serious Adverse Events (participants affected / at risk) | 2/15 | 21/40
Other Adverse Events (participants affected / at risk) | 12/15 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=15) | GDC-0449 (N=40)
Cardiac stent for blocked artery (Cardiac disorders) | 1 | 0
Hysterectomy (Reproductive system and breast disorders) | 1 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 2
Weight loss (Metabolism and nutrition disorders) | 0 | 6
Pneumonia (Infections and infestations) | 0 | 2
Reactions to antibiotic (Injury, poisoning and procedural complications) | 0 | 2 — Reactions to antibiotics include ciprofloxacin and Bactrim
Chest pain (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Hip replacement surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee replacement surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Mesenteric cyst (Gastrointestinal disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=15) | GDC-0449 (N=40)
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 40
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 40
Dysgeusia (Gastrointestinal disorders) | 1 | 37
Gastrointestinal upset (Gastrointestinal disorders) | 2 | 26
Weight loss (Metabolism and nutrition disorders) | 1 | 25
Fatigue (General disorders) | 0 | 19
Common cold (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Acne (Skin and subcutaneous tissue disorders) | 2 | 7
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 5
Dizziness (Vascular disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes